CLINICAL TRIAL: NCT01552135
Title: Pilot Study - Does Nanoparticles in Sunscreen Penetrate Intact or Sunburned Skin?
Brief Title: Pilot Study - Putative Penetration of Nanoparticles in Sunscreen in Intact or Sunburned Skin
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: National Institute of Occupational Health, Norway (Other Government); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Bato Hammarstrøm, MD, Oslo University Hospital
Other Study IDs: 2011/2567B
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Healthy Skin; Sunburned Skin; Titanium Dioxide; Nanoparticles; Penetrate Skin
Keywords: titanium dioxide; nanoparticles; skin; penetrate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy: Healthy men above 50 years old

SUMMARY:
The investigators want to study if nanoparticles of titaniumdioxide are penetrating skin when the skin is intact and when the skin is sunburned. The hypothesis is "Does nanotitandioxide penetrate intact or sunburned skin?"

DETAILED DESCRIPTION:
In this pilotstudy there are two human volunteers. The study comprises two phases. The first phase: The volunteers are applying a commercially available sunscreen lotion containing titanium dioxide nano particles 6 times a day for one week in an area of the back that is 30x20 cm. Before the first application a 2mm punch biopsy is to be taken and examined by scanning electron microscopy. After applying sunscreen lotion for a week, a new biopsy will be taken in order to see how far down in the skin the particles have penetrated. In the second phase: An artificial sunburn will be induced in the same area of the back. They will thereafter apply the sunscreen lotion 6 times a day like in the first phase. After two days (estimated time of maximum skin irritation) a biopsy will be taken in order to see if the nanoparticles have penetrated down in the layers of the skin, and the investigators will also take a biopsy after a full week of applying the sunscreen lotion. The investigators will also examine the urine, before and after the use of sunscreen, to see if the investigators can find the particles there.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men above 50 years old

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2 healthy males older than 50 years
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Depth of penetration of nano particles in skin | One Week

SECONDARY OUTCOMES:
Occurrence of nano particles in urine | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marit Gulbrandsen, MD, Principal Investigator — University Hospital of North Norway; Jan-Oivind Holm, MD PhD, Principal Investigator — Oslo University Hospital; Vidar Skaug, MD, Principal Investigator — National Institute of Occupational Health, Norway; Elise Naess, MD, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Dept. of Environmental and Occupational Medicine, Oslo, Norway